CLINICAL TRIAL: NCT02102867
Title: Evaluating User Perceptions and Experiences of Dual Compartment Microbicide Formulations. Project 5.1: Developing Rectal USPE Measures
Brief Title: Developing Rectal USPE Measures
Acronym: Project DRUM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: ImQuest Pharmaceuticals, Inc. (Industry); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 11968; U19AI101961 (NIH)
Record Dates: First submitted 2014-03-26; First posted 2014-04-03 (Estimated); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Microbicide Delivery System Perceptibility and Acceptability
Keywords: HIV; STI; Primary Prevention; Topical Microbicides; User Experience; Drug Delivery Systems
MeSH Terms: conditions — Sexually Transmitted Diseases | interventions — Gels; Green Or; Fluid Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Formulations (Other): Gel, Cream, Liquid
  Interventions: Other: Gel; Other: Cream; Other: Liquid

INTERVENTIONS:
Other: Gel — 10mL
  Other Names: Orange
Other: Cream — 10mL
  Other Names: Green
Other: Liquid — 10mL
  Other Names: Yellow

SUMMARY:
The purpose of this study is to: (a) adapt existing vaginal USPE items/instruments for evaluation of similar elements of rectal compartment use; (b) develop these scales using 3 distinct semi-solid formulations that represent a range of physicochemical and rheological properties of microbicides that are currently being designed for dual compartment use; and (c) develop novel USPE instruments to capture the experience of product use in the context of receptive anal intercourse (RAI) in both male and female cohorts.

DETAILED DESCRIPTION:
HIV prevention is a global public health priority. Providing efficacious prevention methods that have the greatest likelihood of use will have a profound impact on the public's health. Critical to their use is "acceptability." However, current conceptualizations of adherence and acceptability fail to fully articulate and account for patterns of use and non-use. Formulation properties are critically important to both drug delivery and the user experience. Microbicide developers thus have the opportunity to directly control a formulation's impact on acceptability and adherence to product use, as well as biological product performance. Microbicide products can and should be developed such that they achieve performance standards for both these behavioral (user experience) and biological (efficacy) functions. By incorporating the user experience early on in the product development process, developers will have the greatest chance of providing at-risk individuals with the best prevention methods science can provide. Developing prevention products that can be used in the vagina and/or the rectum and that optimize the user experience in both compartments increases the likelihood that these products will be used consistently and correctly. The impact on global public health has the potential to be far-reaching, decreasing HIV and sexually transmitted infections (STI) incidence and prevalence in both women and men.

Methodology and Data Collection: This is a formative study in which volunteers (N~20-30; ~8-20 males; ~8-20 Females) will first be prescreened for basic study eligibility using a brief questionnaire. Those who are interested in the study and are eligible based on their responses to the prescreen will then complete a STI/HIV screening and pregnancy test (for females).

During the course of the study, participants will evaluate 3 study products (i.e., distinct semi-solid formulations that represent a range of physicochemical and rheological properties). Each participant will be randomly assigned to the order in which they will evaluate the 3 products. After a sexual encounter that includes RAI and study product use, participants will be required to complete a web survey about their experience with the study product.

ELIGIBILITY:
Inclusion Criteria:

* All participants must meet all of the inclusion criteria to participate in this study.

  * Eligible male participants must be 18 years of age or older
  * Eligible female participants must be 18-45 years of age

Inclusion criteria include men and women who:

* Report receptive anal intercourse (RAI) at least twice in the past 6 months,
* Are willing to use each study product in conjunction with RAI on at least one occasion in each data collection period (resulting in a minimum of 3 RAI events during each product evaluation period; on average every 2 weeks, all 3 products across an average of 6 -12 weeks))
* Are willing and able to respond to study data collection systems via phone and internet, attend all study visits, and participate in in-depth qualitative interviews

Exclusion Criteria:

* Male and female participants will be ineligible if they:

  * Have a sensitivity or allergy to vaginal, anal, or rectal products,
  * Have a sensitivity or allergy to any of the ingredients contained in the study products,
  * Are HIV positive at baseline, or have a known HIV-positive sexual partner,
  * Have an active rectal or reproductive tract infection requiring treatment per current Centers for Disease Control (CDC) guidelines or symptomatic urinary tract infection (UTI). Infections requiring treatment include Chlamydia (CT)*, gonorrhea (GC)*, syphilis, active herpes simplex virus (HSV) lesions (note: HSV seropositivity with no active genital lesions is not an exclusion criterion, since treatment is not required), chancroid, genital sores or ulcers, and, if clinically indicated, genital warts,
  * Have current inflammatory bowel disease (IBD) or history of active IBD within last 3 months,
  * Have any other significant colorectal symptom(s) as determined by medical history, participant self-report , or physical exam (including but not limited to presence of any unresolved injury, infectious or inflammatory condition of the local mucosa, presence of symptomatic external hemorrhoids, and presence of any painful anorectal conditions that would be tender to manipulation),
  * Have a nontreatable sexually transmitted disease that could, in the opinion of the investigator/study clinician, make the patient unsuitable for the study or unable to comply with study requirements
  * Have any other clinical condition or prior therapy that, in the opinion of the investigator/study clinician, would make the patient unsuitable for the study or unable to comply with the study requirements,
  * Are unwilling to refrain from use of nonoxynol-9 (N9) for the duration of the study,
  * Are unable or unwilling to communicate in English, or
  * Are unable or unwilling to give written informed consent.

Additionally, female participants will be ineligible if they:

• Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2015-03 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Morrow, PhD, Principal Investigator — The Miriam Hospital: Centers for Behavioral & Preventive Medicine; Robert Buckheit, PhD, Principal Investigator — ImQuest Pharmaceuticals, Inc.
Locations (1):
- The Miriam Hospital: Centers for Behavioral & Preventive Medicine, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited (RI, MA USA) via call-lists, flyers, ads, internet/social media, clinics, CBOs, word-of-mouth.
Pre-assignment Details: Three female participants were withdrawn from study and did not complete product evaluation. One had a positive pregnancy, two withdrew due to not being able to follow study guidelines.
Groups:
- Females: Female participants that reported user sensory perception experiences for 3 formulations (Gel, Cream, and Liquid) during Receptive Anal Intercourse (RAI).
- Males: Male participants that reported user sensory perception experiences for 3 formulations (Gel, Cream, and Liquid) during Receptive Anal Intercourse (RAI).
Period: Overall Study
Arm/Group | Females | Males
Started | 10 | 8
Orange/Gel Use | 7 | 8
Green/Cream Use | 7 | 8
Yellow/Liquid Use | 7 | 8
Completed | 7 (7 pts used all three products (Orange/Gel, Green/Cream, and Yellow/Liquid)) | 8 (8 pts used all three products (Orange/Gel, Green/Cream, and Yellow/Liquid))
Not Completed | 3 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Females: Female participants evaluating three formulations
- Males: Male participants evaluating three formulations
- Total: Total of all reporting groups
Arm/Group | Females | Males | Total
Number analyzed (Participants) | 7 | 8 | 15
Age, Customized [Count of Participants; unit: Participants]
  18-29 Years | 4 | 5 | 9
  30+ Years | 3 | 3 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 0 | 7
  Male | 0 | 8 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black | 3 | 0 | 3
  White | 4 | 7 | 11
  Asian | 0 | 0 | 0
  American Indian/Alaska Native | 0 | 0 | 0
  Hispanic/Latinx | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 8 | 15
Yearly Income [Count of Participants; unit: Participants]
  Less than $15,000 | 2 | 4 | 6
  $15,000-$36,000 | 2 | 3 | 5
  Mora than $36,000 | 3 | 1 | 4
History of STD Diagnosis [Count of Participants; unit: Participants] | 1 | 2 | 3
Vaginal Deliveries [Count of Participants; unit: Participants] — Population: Vaginal deliveries does not apply to Male participants
  Participants
    number analyzed (Participants) | 7 | 0 | 7
    (all) | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: User Sensory Perception & Experience (USPE; Perceptibility) Scale Item Means
Description: USPE Sum of averaged item means/# items (min:max 1:5); 1=Do not agree at all;2=Agree a little;3=Agree somewhat;4=Agree a lot;5=Agree completely.
  Products:Gel/Orange, Cream/Green, Liquid/Yellow. Initial Penetration:Smoothness/lubricity; Initial Lubrication:Coating/lubricating; Spreading Behavior:Ease of stroke, product spread; Product Awareness:Feel during sex (movement, felt betw rectal wall-penis); Perceived Wetness:Covering entire rectum, as after orgasm; Stimulating: enhanced pleasure; Messiness:Perceptions of messiness; Leakage:Sensations of leaking during/after sex, in pubic hair, cleanliness; Pre-coital Leakage:Product felt/leakage on body/clothes before sex; Naturalness:Sensation of naturalness, leakage looked like cum; Lubricity:Wetness before sex; slipperiness/lubricity during sex; Effortful:Effort needed at penetration; effort difficulty/dryness; Pleasure: Partner's stimulation; Noticeable: messiness, thickness
  Higher scores=greater agreement re:product characteristics
Time Frame: 3 web-based surveys over an average of 6-12 weeks
Population: Numbers analyzed for each scale may differ from overall sample size as a function of sex (and hence opportunity to evaluate) or a non-evaluable scale for a given participant.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Females: Female participants that reported user sensory perception experiences for 3 formulations.
- Males: Male participants that reported user sensory perception experiences for 3 formulations.
Arm/Group | Females | Males
Number analyzed (Participants) | 7 | 8
units on a scale
  SEX: Initial Penetration (Green) | 3.67 (1.11) | 3.29 (1.71)
  SEX: Initial Penetration (Orange) | 3.86 (1.35) | 3.42 (1.32)
  SEX: Initial Penetration (Yellow) | 3.86 (0.90) | 3.50 (1.05)
  SEX: Initial Lubrication (Green) | 4.03 (0.78) | 3.15 (1.81)
  SEX: Initial Lubrication (Orange) | 3.74 (0.96) | 3.78 (1.06)
  SEX: Initial Lubrication (Yellow) | 4.17 (0.55) | 3.23 (1.44)
  SEX: Spreading Behavior (Green) | 3.62 (1.22) | 3.25 (1.19)
  SEX: Spreading Behavior (Orange) | 3.48 (1.00) | 3.50 (1.11)
  SEX: Spreading Behavior (Yellow) | 3.62 (0.93) | 3.17 (1.30)
  SEX: Messiness (Green) | 2.71 (0.76) | 1.96 (0.81)
  SEX: Messiness (Orange) | 2.19 (0.72) | 1.79 (0.86)
  SEX: Messiness (Yellow) | 2.40 (1.04) | 2.74 (1.38)
  SEX: Perceived Wetness (Green): number analyzed (Participants) | 7 | 7
  SEX: Perceived Wetness (Green) | 3.68 (1.12) | 2.82 (1.40)
  SEX: Perceived Wetness (Orange) | 3.36 (1.06) | 3.44 (1.18)
  SEX: Perceived Wetness (Yellow): number analyzed (Participants) | 7 | 7
  SEX: Perceived Wetness (Yellow) | 3.43 (0.59) | 2.43 (0.64)
  SEX: Product Awareness (Green): number analyzed (Participants) | 6 | 8
  SEX: Product Awareness (Green) | 3.74 (0.97) | 3.20 (1.14)
  SEX: Product Awareness (Orange) | 3.84 (0.91) | 2.89 (0.99)
  SEX: Product Awareness (Yellow) | 3.73 (0.61) | 3.38 (1.23)
  SEX: Leakage (Green) | 2.86 (1.53) | 2.56 (1.15)
  SEX: Leakage (Orange) | 2.54 (0.64) | 2.34 (0.84)
  SEX: Leakage (Yellow) | 3.11 (0.97) | 3.00 (1.30)
  SEX: Stimulating (Green): number analyzed (Participants) | 6 | 7
  SEX: Stimulating (Green) | 2.86 (1.32) | 2.24 (0.93)
  SEX: Stimulating (Orange) | 2.83 (0.63) | 2.71 (1.24)
  SEX: Stimulating (Yellow): number analyzed (Participants) | 7 | 7
  SEX: Stimulating (Yellow) | 3.00 (0.57) | 2.52 (1.36)
  SEX: Naturalness (Green): number analyzed (Participants) | 7 | 7
  SEX: Naturalness (Green) | 2.43 (0.51) | 2.18 (0.76)
  SEX: Naturalness (Orange) | 2.36 (0.73) | 2.75 (1.21)
  SEX: Naturalness (Yellow) | 2.64 (0.43) | 2.34 (1.00)
  SEX: Lubricity (Green) | 3.52 (1.23) | 2.50 (0.91)
  SEX: Lubricity (Orange) | 3.95 (0.56) | 3.13 (0.94)
  SEX: Lubricity (Yellow): number analyzed (Participants) | 7 | 7
  SEX: Lubricity (Yellow) | 3.48 (0.86) | 3.19 (1.30)
  SEX: Effortful (Green) | 1.50 (0.58) | 1.69 (1.17)
  SEX: Effortful (Orange) | 1.43 (1.13) | 1.97 (1.28)
  SEX: Effortful (Yellow) | 1.36 (0.48) | 1.59 (0.67)
  SEX: Pleasure (Green) | 3.24 (1.58) | 2.96 (1.79)
  SEX: Pleasure (Orange) | 3.62 (1.03) | 2.83 (1.23)
  SEX: Pleasure (Yellow) | 3.52 (0.96) | 2.33 (0.98)
  SEX: Pre-Coital Leakage (Green): number analyzed (Participants) | 4 | 6
  SEX: Pre-Coital Leakage (Green) | 1.67 (0.61) | 1.33 (0.67)
  SEX: Pre-Coital Leakage (Orange): number analyzed (Participants) | 4 | 6
  SEX: Pre-Coital Leakage (Orange) | 1.75 (1.10) | 1.33 (0.67)
  SEX: Pre-Coital Leakage (Yellow): number analyzed (Participants) | 1 | 5
  SEX: Pre-Coital Leakage (Yellow) | 2.00 | 1.87 (1.26)
  SEX: Noticeable (Green) | 3.10 (1.30) | 2.79 (1.15)
  SEX: Noticeable (Orange) | 2.85 (1.00) | 2.63 (1.05)
  SEX: Noticeable (Yellow) | 2.90 (0.74) | 2.25 (0.89)

ADVERSE EVENTS:
Time Frame: 6-12 weeks
Description: Adverse events are combined across arms (Gel/Orange, Cream/Green, Liquid/Yellow) and separated by sex only, since only 1 adverse event with the Cream/Green product was reported overall (female, Cream/Green).
Groups:
- Females: Female participants evaluating three formulations: Gel/Orange; Cream/Green; Liquid/Yellow
- Males: Male participants evaluating three formulations: Gel/Orange; Cream/Green; Liquid/Yellow
Arm/Group | Females | Males
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8
Other Adverse Events (participants affected / at risk) | 1/7 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Females (N=7) | Males (N=8)
Anorectal pain (Green) (Gastrointestinal disorders) | 1 (1) | 0 (0) — Pt reported pain, described as "bloating" when using the cream/green product. It felt like a "glob" of product being pushed further into her rectum during anal sex. Pt evacuated the cream/green product after sex by moving her bowels. Felt fine after.

LIMITATIONS AND CAVEATS:
User Sensory Perceptions & Experience (USPE) scales adapted and were used for the first time to evaluate products used by males for receptive anal sex and females for receptive anal sex.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No